CLINICAL TRIAL: NCT03091387
Title: Utility of Spontaneous Breathing Trial (SBT) Using ET-CPAP, in Predicting Extubation Failure in Neonates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ali S. Hussain, Senior instructor, Aga Khan University
Other Study IDs: SBT NICU
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Neonates
Keywords: neonates, extubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spontaneous Breathing Test — subjects when ready for extubation will be given a three minute spontaneous breathing test on ET-Cpap mode of the ventilator

SUMMARY:
Intubation and ventilation are lifesaving interventions in the neonatal intensive care unit (ICU), especially among preterm, low birth weight babies. However, timely extubation is also necessary. The decision to extubate usually depends on clinical judgement, appropriate blood gas prior to extubation and low ventilator parameters. Approximately 40 % of babies' extubated on the above criteria require re-intubation, suggesting that current methods to predict extubation failure are insufficient. . Spontaneous breathing trial (SBT) has been predominantly used in infants and children to access the readiness for extubation. Few studies in premature neonates have also shown good sensitivity and specificity in predicting extubation success. However its significance in our population is yet to be determined. We aim to use this for both our preterm and term babies and if results are significant we plan to include this as our routine pre extubation criteria.

DETAILED DESCRIPTION:
Intubation and ventilation are lifesaving interventions in the neonatal intensive care unit (ICU), especially among preterm, low birth weight babies. However, timely extubation is also necessary, in order to prevent adverse effects of prolonged intubation, such as iatrogenic pneumothorax, superadded bacterial infections and colonization, subglottic injury and bronchopulmonary dysplasia1,2.

For extubation to be successful, baby should maintain hemodynamic stability and O2 saturation for at least 48 hours post-extubation. So far there are no standard guidelines, especially in low resource countries such as ours, to predict successful extubation. The decision to extubate usually depends on clinical judgement, appropriate blood gas prior to extubation and low ventilator parameters3. Intensivists may vary in their experience and training, resulting in a large variation in the timing and outcome of extubation.

Research from high income settings indicates that approximately 40 % of babies extubated on the above criteria require re-intubation, suggesting that current methods to predict extubation failure are insufficient.3 Readiness for extubation can be objectively measured by observing pulmonary functions, respiratory muscle strength, respiratory drive, ventilator flow volumes and gas exchange.5,6 Re-intubation causes prolonged hospital stay, adversely effects the family, and results in undesirable effects on the neonate4 . Therefore accurate prediction of extubation failure in neonates is a high priority. Spontaneous breathing trial (SBT) has been predominantly used in infant and children to access the readiness for extubation . Few studies in premature neonates have also shown good sensitivity and specificity in predicting extubation sucess7.However its significance in our population is yet to be determined. We aim to use this for both our preterm and term babies and if results are significant we plan to include this as our routine pre extubation criteria.

Primary Objective:

To evaluate the usefulness of SBT, in predicting extubation failure among neonates admitted to a NICU in a tertiary care hospital in Karachi, Pakistan.

Secondary Objective:

1. To evaluate the usefulness of ratio of spontaneous expired minute ventilation(VE) during ET CPAP to VE during mechanical ventilation (V˙E ratio , )in predicting extubation failure among neonates admitted to a NICU in a tertiary care hospital in Karachi, Pakistan.
2. To evaluate the usefulness of VE during ETCPAP, in predicting extubation failure among neonates admitted to a NICU in a tertiary care hospital in Karachi, Pakistan.

Study Design: Prospective validation study Study Setting: NICU, AKU Duration of study: 12 months Study Population: Neonates admitted to a tertiary care NICU in a low resource setting

Operational definitions:

1. Expired Tidal volume(Vte) : volume of gas (ml) which moves out of the lung with each breath.
2. Spontaneous Expired Minute ventilation(VE) : amount of gas spontaneously exhaled from lungs in one minute. This is a product of Vte and respiratory rate. It is displayed in real time on SLE 5000 ventilator. Normal values for full term babies is 200-400 ml/kg/min whereas 200-300 ml /kg/min for preterm babies.
3. VE Ratio: Et cpapVE/Vent VE Sampling technique: Consecutive sampling Sample size: Assuming SBT to have 95% sensitivity and 73% specificity for predicting extubation sucess7 , and presuming that 30% of neonates will fail extubation, we will require 45 neonates in each group to obtain 95% CIs of ±3%. The sample size will be inflated by 20% to accommodate for differences in re-intubation practice. Therefore 55 neonates in each group will be enrolled in the study. This sample size is sufficient to also detect a difference of 1 SD in mean VE in the group failing extubation, assuming an overall mean VE of 300ml/kg/min (power 80%and twotail αof 0.05).

Study Methods:

Identification and recruitment of neonates:

An NICU fellow not involved in the clinical management of the baby will maintain a log of all neonates who are planned to be extubated. Eligibility assessment will be done by the fellow who will then approach the neonate's family for consent. Care will be taken to ensure that consent is voluntary. Refusal of consent will not lead to any change in the management. A baseline questionnaire will be filled, including demographic information such as post -natal age, gender, gestational age, current weight etc. Information related to the clinical indication of extubation, other medications given will be recorded. Eligible candidates will be divided into two groups of <1.5kg weight and >1.5kg weight. Separate log will be maintained for both groups. Total of 55 enrolments will be made in each group.

Data collection:

Will be according to SOP. Questionnaires are attached.

Index Maneuver:

After enrolment, Nicu SBT study fellow will observe and record clinical data and patient demographics on a predefined proforma. Vitals, including heart rate, respiratory rate, ventilator parameters and respiratory volumes will be recorded by same observer for 3 minutes at 30 second intervals.

After 3 minutes the baby will be shifted to ET CPAP mode on the same ventilator and the same parameters will be rerecorded at 30 sec interval for 3 minutes as done previously. A regularly serviced and authorized stop watch will be used to monitor the time and all parameters will be recorded from the Mindray (IPM12) monitors and SLE 5000 ventilator. The clinical teams caring for the patients will not be present during the maneuver and all the babies will be extubated as per the primary teams plan.

Criteria for stopping the index maneuver:

Bradycardia (Heart rate <100bpm) for >15 seconds and/or oxygen Saturation of <85% even after 15 % increase in Fi02 from the baseline.

Follow-up and outcomes:

Outcomes of extubation will be recorded separately after 48 hours. The reasons for re-intubation will also be recorded.

Blinding:

SBT maneuver will be performed by a fellow not involved in the clinical team. The clinical team will be blinded to the results of the SBT. The success and failure of SBT will be determined by the principal investigator, who will be blinded to the outcome of the extubation, after the completion of the study

SBT Results: SBT will be labeled as failed if the criteria for stopping the index maneuver were applied.

Analysis plan:

Descriptive analysis for both groups will be performed for continuous variables like age, weight , gestational age , chronological age using means with SD and medians with interquartile ranges as appropriate. For categorical variables e.g. gender, frequencies and proportions will be reported. Multiple logistic regression will be done to identify factors predicting SBT failure in each group. P value of < 0.05 will be taken as significant..

Sensitivity, specificity, PPV, NPV, LR will be calculated using area under curve (AUC).

Subgroup analysis for secondary outcomes will be performed in different gestational age and weight categories.

Continuous outcomes will be compared using student's t test when normally distributed and by Mann-whitney U test when skewed. Categorical data will be assessed using the chi square test and fisher two tailed exact test where indicated. The ability of the outcome (SBT, VE, VE ratio) variables to accurately discriminate between successful and failed extubation will be assessed using receiver operating curves(ROC) .

ETHICAL CONSIDERATIONS

Informed Consent The informed consent will be confirmed with a signature or thumbprint by the parent or the authorized guardian of the child. In the absence of a signature, a witness (other than the member of the research team obtaining consent) will be asked to sign. Finally, the member of the research team obtaining consent will sign this form.

Safety and Risks There is a potential risk of transient hemodynamic instability when performing the SBT. That is why, safety net is in place to record heart rate and O2 saturation every 30 seconds. A trained nurse and neonatal fellow trained in NRP will be available at the bedside during the procedure. The fellow performing the procedure is year two with NRP certification. He will further be trained to immediately revert to the ventilation mode if HR < 100 beats per minute for > 15 seconds and increase in Oxygen requirement O2. This has been practiced in another study in an NICU by PG Davis et al in 2006 and shown to have no adverse effects7.

Vulnerable Populations Study population is neonates because the study involves optimizing NICU care of neonates. Consent will be taken in Urdu to ensure that the potential participant understands the research. Extra protection will be in place to ensure voluntary participation. It will be explained that participation is voluntary and can be terminated by the participant at any time without reason and without any penalty. If the potential participant has any questions, they will be answered in their native language to ensure that they understand the research and their potential role in it. The study personnel will not influence the clinical team's decisions in caring for the neonate.

Confidentiality To ensure privacy, all the interviews will take place in a separate room. Hard copies of the study-related forms will be stored in a locked cabinet in a storage room under supervision of the principal investigators. Only approved study personnel will have access to this information. After completion of the study, identifier information will be stripped and only study IDs will be used during analysis. All identifier information will be delinked and identifier information will be stored under lock and key.

ELIGIBILITY:
Inclusion Criteria:

* 1. Neonates who are intubated for more than 24 hrs. AND 2. Extubation is planned by the primary team onto Nasal continuous positive airway pressure (NCPAP) for weight < 1.5 kg OR Oxygen via nasal prongs for weight ≥ 1.5 kg

AND having all of the following:

1. Pre extubation blood gas pH=7.25-7.45 and PCo2=35-45mmHg
2. Pre extubation fractional inspiration of oxygen (FiO2)=<40%
3. Is off sedation medication for >4 hrs
4. I-time= 0.3-0.36 sec
5. Peep: 5 cm h20
6. VTe: >3 ml/kg
7. Breathing rate above the set ventilator rate

   4. Family providing written informed consent

   Exclusion Criteria:
   1. Neonates who will be extubated and kept on other modalities like high flow nasal cannula.
   2. Congenital malformation like lung hypoplasia/diaphrgmatic hernia/congenital cyanotic heart disease.
   3. Neonate with suspicion of neuromuscular disorder.
   4. Neonates with accidental extubation

      -

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates on mechanical ventilation in NICU.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | 48hrs
  reintubation within 48 hrs of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Ali S. Hussain, MBBS,FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bancalari E, Sinclair J. Effective care of the newborn infant, 1st ed. New York: Oxford University Press, 1992.
- [Background] Halliday HL. Towards earlier neonatal extubation. Lancet. 2000 Jun 17;355(9221):2091-2. doi: 10.1016/s0140-6736(00)02372-2. No abstract available. PMID 10902619
- [Background] Stefanescu BM, Murphy WP, Hansell BJ, Fuloria M, Morgan TM, Aschner JL. A randomized, controlled trial comparing two different continuous positive airway pressure systems for the successful extubation of extremely low birth weight infants. Pediatrics. 2003 Nov;112(5):1031-8. doi: 10.1542/peds.112.5.1031. PMID 14595042
- [Background] Fox WW, Schwartz JG, Shaffer TH. Successful extubation of neonates: clinical and physiological factors. Crit Care Med. 1981 Dec;9(12):823-6. doi: 10.1097/00003246-198112000-00003. PMID 7318452
- [Background] Khan N, Brown A, Venkataraman ST. Predictors of extubation success and failure in mechanically ventilated infants and children. Crit Care Med. 1996 Sep;24(9):1568-79. doi: 10.1097/00003246-199609000-00023. PMID 8797633
- [Background] Baumeister BL, el-Khatib M, Smith PG, Blumer JL. Evaluation of predictors of weaning from mechanical ventilation in pediatric patients. Pediatr Pulmonol. 1997 Nov;24(5):344-52. doi: 10.1002/(sici)1099-0496(199711)24:53.0.co;2-i. PMID 9407568
- [Background] Kamlin CO, Davis PG, Morley CJ. Predicting successful extubation of very low birthweight infants. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F180-3. doi: 10.1136/adc.2005.081083. Epub 2006 Jan 12. PMID 16410255